CLINICAL TRIAL: NCT05276011
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Determine the Efficacy, Safety, and Dosing of TG-C in Adult Subjects with Symptomatic Early Hip Osteoarthritis
Brief Title: A Study to Determine the Safety and Efficacy of TG-C in Subjects with Symptomatic Early Hip Osteoarthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kolon TissueGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGC-OAH-201
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Osteoarthritis
Keywords: hip
MeSH Terms: conditions — Joint Diseases | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Treatment (TG-C) (Active Comparator): TG-C at 1.0 x 10e7 cells per single 2 mL intraarticular injection
  Interventions: Biological: TG-C
- Active Treatment 2 (TG-C) (Active Comparator): TG-C at 3.0 x 10e6 cells per single 2 mL intraarticular injection
  Interventions: Biological: TG-C
- Placebo Control (Normal Saline) (Placebo Comparator): Normal saline, single 2 mL intraarticular injection
  Interventions: Biological: Placebo Control

INTERVENTIONS:
Biological: TG-C — 2 mL injection of non-transduced human chondrocytes and irradiated transduced human GP2-293 cells expressing TGF-B1.
  Other Names: TissueGene-C
  Arms: Active Treatment (TG-C); Active Treatment 2 (TG-C)
Biological: Placebo Control — 2 mL normal saline injection
  Other Names: Normal Saline
  Arms: Placebo Control (Normal Saline)

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Determine the Efficacy, Safety, and Dosing of TG-C in Adult Subjects with Symptomatic Early Hip Osteoarthritis. TG-C will be administered to the target hip by a single ultrasound (or fluoroscopy)-guided, intra-articular injection with image capture showing correct injection of study drug into the femoroacetabular joint. Patients will be followed for 12 months for safety and efficacy.

DETAILED DESCRIPTION:
This protocol is designed to assess the safety and efficacy of TG-C in treating symptoms of osteoarthritis of the hip and determining disease modifying effects of TG-C. TG-C will be compared to normal saline as a control. Safety will be evaluated by observation of the injection site for irritation or other effects, the incidence and severity of adverse events, and changes in physical examination findings, radiographic criteria, and laboratory tests. Patients will be followed for 12 months for both safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years old
* The subject has a diagnosis of Grade ≤2 primary OA of the target hip
* Pain ≥ 40 on VAS scale
* The subject has groin pain that is elicited by hip rotation on physical examination
* No history of significant organ system disorders.
* Body mass index (BMI) <40 kg/m2
* Systolic blood pressure of 100 to 160 mmHg and diastolic blood pressure of 60 to 90 mmHg.
* Using birth control
* Written informed consent

Exclusion Criteria:

* The subject exhibits severe symptoms in the target hip that result in difficulty or an inability to walk.
* The subject has severe hip OA ipsilateral to the target hip.
* Previous cartilage transplantation procedure to the injured cartilage surface.
* Major injury to the target hip within 12 months of screening.
* Active dermal ulcer or infection in the proximity of the target hip within 1 month before screening.
* The subject has had surgery on the target hip within the last 6 months.
* Total hip replacement surgery or other surgery on the target hip in the next 12 months.
* MRI indicates bone marrow infiltration, fracture, osteonecrosis/bone infarct, osteochondritis dissecans, tumor, moderate to severe dysplasia, avascular necrosis, post-traumatic arthritis, transient osteoporosis, slipped-cap femoral epiphysis, juvenile idiopathic arthritis, or axial juvenile spondyloarthritis.
* Hip conditions including but not limited to any autoimmune or infectious cause for arthritis; metabolic joint disease; neuropathic disorders, groin pain from non-orthopedic sources, or tumors, congestive heart failure, or chronic kidney disease.
* Uncontrolled diabetes based on a hemoglobin A1c (HbA1c) value >8% at the screening Visit.
* Increased risk for post-procedure bleeding or post-procedure infection.
* Ongoing infectious disease, including, but not limited to, HIV, hepatitis C, or current or prior hepatitis B.
* Cognitive impairment that would limit his/her ability to provide informed consent or to complete assessments and questionnaires.
* 1 year history of drug or alcohol abuse.
* Contraindication to or cannot undergo MRI.
* Active malignancy within the last 5 years.
* Pregnant or is lactating.
* Taken steroidal or NSAIDs within 14 days before the Baseline Visit
* Using topical analgesics on the target hip
* Receiving chronic narcotic treatment at screening.
* Received any injection to the target hip within the 3 months before the Baseline Visit.
* Taking antiplatelet or anticoagulants.
* Participated in an investigational study within 13 weeks before the Screening Visit or in the next 25 months.
* Unable to comply with the requisite study follow-up and all of the follow-up office visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Hip Pain as Assessed by VAS | Baseline to Month 12
  Assessment of change from baseline in target hip pain using the Visual Analog Scale (VAS). The VAS is a method for the assessment of the intensity of pain. The VAS is a horizontal line, 100 mm in length and anchored by word descriptors at each end (no pain, very severe pain). The patient marks on the line at the point that represents their current state. The VAS score is determined by measuring in millimeters from the left hand end to the point of the mark. The score ranges from "0" or no pain to "100" very severe pain.

SECONDARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score (HOOS) | Baseline to Month 12
  The HOOS questionnaire was built upon the Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC®). Questions from the WOMAC® were used as the basis for the survey, and 2 dimensions were added: sport and recreation and hip-related quality of life. The HOOS is composed of 40 questions in 5 subscales: Pain (10 items), Symptoms (5 items), Activity of Daily Living (17 items), Sport and Recreation Function (4 items), and Hip-Related Quality of Life (4 items). A total score, ranging from 0 to 100 is calculated. Higher scores represent better functioning.
Timed Up and Go Test (TUG) | Baseline to Months 1, 3, 6, 9, and 12
  The TUG test is used to determine the time needed to progress from sitting to standing and walking. In addition, the test helps to evaluate the probability for falls. The individual starts in a seated position in a chair with armrests and, upon command, stands up, walks 3 meters, turns around, walks back to the chair, and sits down. The time stops when the subject is seated. The use of walking aids should be recorded and kept consistent between tests.
UCLA Activity Score | Baseline to Months 1, 3, 6, 9, and 12
  The UCLA Activity Score includes 10 statements that cover the range of activity states from being "wholly inactive, dependent on others, and cannot leave residence" to "regularly participate in impact sports." The respondents are instructed to select one statement that is most representative of their current activity. Lower scores on the scale reflect a low level of activity and higher scores reflect more activity.
Joint Space Width (JSW) on standing X-ray | Baseline to Month 12
  To evaluate the effects of 2 dose levels of TG-C on the structural features of the hip joint
WOMAC® (Western Ontario and McMaster Universities Osteoarthritis Index) total score | Baseline to Month 12
  To evaluate the effects of 2 dose levels of TG-C on symptoms of OA of the hip. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

OTHER OUTCOMES:
Physical Component Score (PCS) of the Short Form 12-Item Health Survey (SF-12 Questionnaire) | 12 months
  Evaluation the Health-Related Quality of Life (HRQoL) as measured by the physical component score (PCS) of the 12-Item Short-Form Health Survey version 2 (SF-12v2®) questionnaire addresses physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. The mean score is set to 50. Scores >50 indicate better physical or mental health than the mean, and scores <50 indicate worse physical or mental health than the mean.
Clinician Global Impression of Change (CGI-C) | Week 1 and Months 1, 3, 6, 9, and 12
  The CGI-C asks clinicians to choose the response that best describes the overall change in the patient's OA since they received the study medication as "much better," "moderately better," "a little better," "no change," "a little worse," "moderately worse," or" much worse." Clinicians are also asked to indicate if the change that the patient has experienced is clinically meaningful.
Clinician Global Impression of Severity (CGI-S) | Baseline and at Months 1, 3, 6, 9, and 12
  clinician to choose the response that best describes the severity of the patient's overall OA as "none," "mild," "moderate," or "severe."
Patient Global Impression of Severity (PGI-S) | Baseline and at Months 1, 3, 6, 9, and 12
  patients to select the response that best describes the severity of their OA, their OA-related pain, and their OA-related stiffness and their difficulty with activities as a result of their OA as "none," "mild," "moderate," or "severe."
Patient Global Impression of Change (PGI-C) | Week 1 and Months 1, 3, 6, 9, and 12
  patients to choose the response that best describes the overall change in their OA, their OA-related pain, and their OA-related stiffness and the change in their difficulty with activities as a result of their OA since they received the study medication as "much better," "moderately better," "a little better," "no change," "a little worse," "moderately worse," or "much worse." Patients are also asked to indicate if the change that they have experienced is meaningful to them ("yes," "no," or "not applicable" in the case of no change)

CONTACTS AND LOCATIONS:
Overall Officials: Moon Jong Noh, PhD, Study Chair — Kolon TissueGene, Inc.

IPD SHARING:
Plan to Share IPD: No